CLINICAL TRIAL: NCT03056768
Title: Taiwan Health Promotion Intervention Study for Elders
Acronym: THISCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Principal investigator, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14001A
Record Dates: First submitted 2017-02-02; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Frail Elderly Syndrome; Cognitive Impairment; Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active control (Active Comparator): Health promotion provided by local health bureau.
  Interventions: Behavioral: Active control
- multidomain intervention (Experimental): 1-year multidomain health promotion (physical activities, cognitive training, nutritional sessions)
  Interventions: Behavioral: Multidomain intervention

INTERVENTIONS:
Behavioral: Multidomain intervention — 1-year multidomain health promotion (physical, cognitive, nutritional intervention)
  Arms: multidomain intervention
Behavioral: Active control — Health promotion activities provided by local health bureau.
  Arms: active control

SUMMARY:
Objectives: 1-year multidomain health promotion on prevention of physical and cognitive decline for community-living older people.

Design:

Methods: Randomized controlled trial

Setting:

Five cities(Taipei, Taichung, Kaohsiung, Kinmen, I-Lan) in Taiwan Participants: age 65 or older community-dwelling prefrail or frail adults Intervention: 1-year multidomain health promotion (physical, cognitive, nutritional intervention)

Measurements:

Primary outcome includes frailty status and cognitive performance. Secondary outcomes include depressive symptoms, nutrition assessment, and functional capacity; All the variables were measured at 0, 6, 12 months. The effect of intervention was investigated by intention-to-treat analysis.

DETAILED DESCRIPTION:
Eligibility criteria includes: community-dwelling older people aged 65 or older, and those with confirmed diagnosis of dementia or dependent on activities of daily living were excluded.

Primary outcome includes frailty status measured by CHS frailty score. general and sub-domain cognitive performance measured by Montreal Cognitive Assessment (MoCA). Secondary outcomes include depressive symptoms, nutrition assessment, and functional capacity; which were evaluated by 5-item Geriatric Depression scale(GDS-5), Mini-nutrition Assessment(MNA), and instrumental activities of daily living (IADL) individually.

ELIGIBILITY:
Inclusion Criteria:

* Prefrail or frail community-dwelling people

Exclusion Criteria:

* Institutionalized or ADL dependent
* Diagnosed dementia
* Limited life expectancy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1080 (Actual)
Dates: Start 2014-08-30 (Actual); Primary Completion 2015-10-05 (Actual); Study Completion 2016-07-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline frailty score at 12 months | 12 months
  Measured by Cardiovascular Health Study(CHS) definition

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Kung Chen, MD, PhD, Principal Investigator — Director, Center for Geriatrics and Gerontology, Taipei Veterans General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho MY, Lee WJ, Yen KH, Liang CK, Peng LN, Lin MH, Loh CH, Hsiao FY, Chen LK. Tailoring multidomain intervention programs to reduce cognitive and physical decline in older adults: Examining rural-urban differences in a nationwide cluster-randomized controlled trial. J Prev Alzheimers Dis. 2025 Sep;12(8):100231. doi: 10.1016/j.tjpad.2025.100231. Epub 2025 Jun 12. PMID 40514302